CLINICAL TRIAL: NCT00003863
Title: Genetic Changes in Diffuse Aggressive Non-Hodgkin's Lymphoma
Brief Title: Diagnostic Study of Patients With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9764; U10CA076001 (NIH); CALGB-9764; CDR0000067027 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult Burkitt lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; stage I mantle cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Comparative Genomic Hybridization; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Gene Rearrangement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Tissue samples are obtained before treatment and at the time of documentation of refractory disease in patients who do not achieve complete remission after induction therapy or at the time of first relapse in patients who achieve a complete remission.
  Samples are examined for rearrangements in the MYC, BCL2, BCL6, and IGH genes using fluorescent in situ hybridization. DNA is examined by comparative genomic hybridization, which allows cytogenetic detection of losses and gains of chromosomal regions in tumor cells.
  Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.
  Interventions: Genetic: comparative genomic hybridization; Genetic: cytogenetic analysis; Genetic: fluorescence in situ hybridization; Genetic: gene rearrangement analysis

INTERVENTIONS:
Genetic: comparative genomic hybridization
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Genetic: gene rearrangement analysis

SUMMARY:
RATIONALE: Determination of genetic markers for aggressive non-Hodgkin's lymphoma may help identify patients with this disease and help predict the outcome of treatment.

PURPOSE: Diagnostic study to determine the genetic markers in patients who have aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the proportions of patients with diffuse aggressive non-Hodgkin's lymphoma who have rearrangements affecting the MYC, BCL2, and BCL6 genes (determined by fluorescent in situ hybridization), overtly amplified chromosomal regions, and nonrandom copy number changes of chromosomal regions (determined by comparative genomic hybridization).
* Investigate the prognostic importance of these genetic markers by studying their relationships with clinical outcomes (e.g., response to therapy, failure-free survival, and overall survival) in these patients.
* Investigate the interrelationships among these genetic and biological markers and their relationships with clinical features of the disease, such as disease site (nodal vs extranodal) and stage, in these patients.

OUTLINE: This is a multicenter study.

Tissue samples are obtained before treatment and at the time of documentation of refractory disease in patients who do not achieve complete remission after induction therapy or at the time of first relapse in patients who achieve a complete remission.

Samples are examined for rearrangements in the MYC, BCL2, BCL6, and IGH genes using fluorescent in situ hybridization. DNA is examined by comparative genomic hybridization, which allows cytogenetic detection of losses and gains of chromosomal regions in tumor cells.

Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven aggressive non-Hodgkin's lymphoma and registered to front-line CALGB protocols (e.g, CLB-59903, 59909, 10002, and 50103)

  * Diffuse small cleaved cell lymphoma
  * Diffuse mixed small and large cell lymphoma
  * Diffuse large cell lymphoma
  * Diffuse large cell immunoblastic lymphoma
  * Small noncleaved cell lymphoma
  * Mantle cell lymphoma OR
* Previously entered on similar curative CALGB protocols (CLB-8852, CLB-8854, and CLB-9351) with blocks or unstained slides of initial diagnosis available

PATIENT CHARACTERISTICS:

Age:

* 18 years and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-Hodgkin's lymphoma and previously enrolled on CALGB 59903, 59909, 10002 and 50103.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 1999-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
response to therapy | Up to 5 years

SECONDARY OUTCOMES:
failure-free survival | Up to 5 years
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Raju Chaganti, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (69):
- United States (69):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Care Center at Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia